CLINICAL TRIAL: NCT07203976
Title: Visual and Refractive Outcomes Following Stream Light Photorefractive Keratectomy (55μm Epithelial Removal) Versus Conventional Photorefractive Keratectomy
Status: Active, not recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Menatallah Gamal Saleh, lecturer of ophthalmology, Assiut University
Other Study IDs: 04-2025-300627
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Photorefractive Keratectomy
Keywords: stream light photorefractive keratectomy; conventional photorefractive keratectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients aged 18-40 years, myopia up to -6.00 D and astigmatism up to -3.00 D and Stable refraction: The visual and refractive outcomes of Stream Light Photorefractive keratectomy with fixed epithelial removal.
- Patients aged 18-40 years, myopia up to -6.00 D and astigmatism up to -3.00 D and Stable refraction: The visual and refractive outcomes of manual Photorefractive keratectomy with fixed epithelial removal.

SUMMARY:
Photorefractive keratectomy (PRK) is a well-established corneal refractive surgery that involves epithelial removal followed by stromal ablation to correct myopia, hyperopia, and astigmatism. The method of epithelial removal in PRK significantly impacts healing, pain levels, and visual outcomes.

Trans-epithelial PRK (StreamLight) performed on the EX500 excimer laser platform removes the epithelium and reshapes the corneal stroma in a single laser-guided step, potentially reducing tissue manipulation and enhancing epithelial healing. In contrast, manual epithelial removal PRK involves mechanical debridement, with epithelial removal depth being manually controlled. The variability of epithelial thickness in StreamLight PRK may influence visual outcomes, whereas in manual PRK, a fixed epithelial removal depth of 55 microns provides a standardized approach.

DETAILED DESCRIPTION:
This study aimed to compare the visual and refractive outcomes of StreamLight PRK versus manual PRK with fixed epithelial removal.

Type of the study: Retrospective cross-sectional study

* Study Setting: Alforsan Eye Centre
* Study subjects:

  a. Inclusion criteria:
  * Patients aged 18-40 years.
  * Myopia up to -6.00 D and astigmatism up to -3.00 D.
  * Stable refraction for at least one year.
  * No history of ocular surgery or corneal pathology. b. Exclusion criteria:
  * Presence of keratoconus or suspected corneal ectasia.
  * Severe dry eye disease or significant ocular surface disease.
  * History of autoimmune disease or systemic conditions affecting wound healing.
  * Prior herpetic eye disease. c. Sample Size Calculation: A sample size calculation will be performed to ensure adequate statistical power. Anticipated enrollment: [e.g., 50 eyes per group] based on previous PRK outcome studies (Marshall et al., 2018).
* Study tools (in detail, e.g., lab methods, instruments,steps, chemicals, …):

  * Alcon Wavelight EX500 excimer laser (Alcon Laboratories, Fort Worth, TX, USA)
  * Wavelight Oculyzer II Am Wolfsmantel 5, Erlangen, Germany
  * Autorefractor KR-8900 (Topcon, Tokyo, Japan)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-40 years.
* Myopia up to -6.00 D and astigmatism up to -3.00 D.
* Stable refraction for at least one year.
* No history of ocular surgery or corneal pathology.

Exclusion Criteria:

* Presence of keratoconus or suspected corneal ectasia.
* Severe dry eye disease or significant ocular surface disease.
* History of autoimmune disease or systemic conditions affecting wound healing.
* Prior herpetic eye disease.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients aged 18-40 years with myopia up to -6.00 D and astigmatism up to -3.00 D and Stable refraction for at least one year.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-03 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Post operative distant uncorrected visual acuity | 1 year
  using snellen chart

SECONDARY OUTCOMES:
Post operative spherical equivalent of refractive error | 1 year
  using autorefractometer

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Assiut, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 3. Marshall, J., Trokel, S. L., Rothery, S., & Krueger, R. R. (2018). Refractive corneal surgery: The role of epithelial healing and biomechanics. Cornea, 37(7), 853-860.
- [Background] Fantes FE, Hanna KD, Waring GO 3rd, Pouliquen Y, Thompson KP, Savoldelli M. Wound healing after excimer laser keratomileusis (photorefractive keratectomy) in monkeys. Arch Ophthalmol. 1990 May;108(5):665-75. doi: 10.1001/archopht.1990.01070070051034. PMID 2334323